CLINICAL TRIAL: NCT02415218
Title: Clinical Study of Transplantation of Autologous Cultivated Oral Mucosal Epithelial Sheets for Limbal Stem-cell Deficiency
Brief Title: Transplantation of Autologous Oral Mucosal Epithelial Sheets for Limbal Stem-cell Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Siriraj Hospital (Other)
Collaborators: Osaka University (Other)
Responsible Party: Principal Investigator, Adisak Wongkajornsilp, M.D., Ph.D., Siriraj Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 662/2555(EC2)
Record Dates: First submitted 2015-04-08; First posted 2015-04-14 (Estimated); Last update posted 2019-10-11 (Actual); Status verified 2019-10

CONDITIONS: Limbal Stem-cell Deficiency
MeSH Terms: conditions — Limbal Stem Cell Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mucosal cell sheet transplantation (Experimental): The subjects will have their oral mucosal tissues retrieved for cell sheet preparation. The mucosal cell sheet will be transplanted over the affected cornea.
  Interventions: Biological: Mucosal cell sheet transplantation

INTERVENTIONS:
Biological: Mucosal cell sheet transplantation — The subjects will have their oral mucosal tissues retrieved for cell sheet preparation. The mucosal cell sheet will be transplanted over the affected cornea.

SUMMARY:
The study purpose is to evaluate the efficacy and safety of cultivated oral mucosal epithelial sheet transplantation as a novel therapy for limbal stem cell deficiency, for which no effective approaches has thus far been available, for the purpose of establishing this therapy as an effective strategy for this disease with an aim of improving visual acuity and corneal transparency.

DETAILED DESCRIPTION:
The efficacy and safety of cultivated oral mucosal epithelial sheet transplantation as a novel therapy for limbal stem-cell deficiency, for which no effective approaches have thus far been available, will be evaluated for the purpose of establishing this therapy as an effective strategy for this disease with an aim of improving visual acuity and corneal transparency. The primary endpoint will be an area of no conjunctivalization and no corneal epithelial defect at one year, which will be evaluated according to a 6-grade rating scale. The secondary endpoints will be corrected visual acuity, severity of corneal opacification, extent of corneal neovascularization, expected ocular complications, and all adverse events including abnormal laboratory findings. The purpose of this research is to evaluate the efficacy of the investigational therapy so as to provide rationales for making this strategy approved as an advanced medical care in the future.

ELIGIBILITY:
Inclusion Criteria:

* Among patients with bilateral limbal stem-cell deficiency, those who meet all the criteria listed below when they give their informed consent to participate in this research will be included.

  1. Patients in whom the eye(s) (subject to the interventional therapy) show(s) loss or dysfunction of corneal epithelial stem cells throughout the total* circumference of the cornea
  2. Patients in whom the corneal surface of the eye(s) (subject to the investigational therapy) is(are) entirely enveloped by conjunctival tissue
  3. Patients of both genders aged ≥20 years when they give their informed consent
  4. Patients who have given their own written consent to participate in this clinical research (The target disease is bilateral limbal stem-cell deficiency, although it is not always necessary that the both eyes of the patient meet the inclusion criteria.)

Exclusion Criteria:

1. Patients who are or may be pregnant, and patients who are breast feeding
2. Patients with infections (HBV, HCV, HIV, HTLV-1)
3. Patients with extreme hypolacrimation resistant to therapy
4. Patients from whom oral mucosal specimens cannot be collected because clear scar formation or inflammatory findings are noted in a cell-collection site of the mucosal membrane
5. Patients whose score of Performance Status (PS*) is 3 or more
6. Any others who are judged by the chief subinvestigator to be ineligible for this clinical research, due to the presence of complications, etc.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-04-17; Primary Completion 2016-09-03 (Actual); Study Completion 2017-04-16 (Actual)

PRIMARY OUTCOMES:
Evaluation of conjunctivalization and corneal epithelial defect | 1 year after transplantation
  One year after the transplantation, an area of no conjunctivalization and no corneal epithelial defect will be rated according to the Grading scale described in Table 2, on the basis of which the efficacy of the investigational therapy will be assessed. Generally, the preoperative condition of ocular surface is rated as "Bad (Grading 0)." In subjects showing improvement to Grading 2 or greater, the investigational therapy will be assessed as effective.

SECONDARY OUTCOMES:
Corrected visual acuity (efficacy) | 1 year
  Corrected visual acuity will be evaluated by the decimal acuity method and converted to Log MAR values, which will be used to assess the extent of postoperative change in visual acuity. Note that 0.005 will be given to "counting fingers," 0.002, to "hand motion," and 0.001, to "light perception" 14). Visual acuity will be measured before transplantation, and 1, 3, and 6 months as well as one year after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Adisak Wongkajornsilp, M.D., Ph.D., Principal Investigator — Mahidol University
Locations (1):
- Siriraj Clinical Research Center, Siriraj Hospital, Bangkoknoi, Bangkok, Thailand

REFERENCES:
- [Derived] Booranapong W, Kosrirukvongs P, Duangsa-Ard S, Kasetsinsombat K, Sa-Ngiamsuntorn K, Wongkajornsilp A. Transplantation of autologous cultivated oral mucosal epithelial sheets for limbal stem cell deficiency at Siriraj Hospital: a case series. J Med Case Rep. 2022 Aug 4;16(1):298. doi: 10.1186/s13256-022-03502-8. PMID 35922868